CLINICAL TRIAL: NCT06308042
Title: Remote Reliability Of 30 Seconds Sit And Stand Test In Patients With Multiple Sclerosis
Brief Title: Remote Evaluation in Patients With Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate professor, physiotherapist,, Inonu University
Other Study IDs: 2024/5558
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: 30 SECONDS SIT AND STAND TEST; REMOTE RELIABILITY
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Acetamido-4'-isothiocyanatostilbene-2,2'-disulfonic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 30 second sit and stand test — The individual sits in the middle of the chair with his back upright, his feet on the ground, and his arms crossed in front of his chest. The individual starts the test with the start command while in this position and takes off as fully as he can for 30 seconds.

SUMMARY:
This study aimed to demonstrate the remote reliability of the 30-second sit-to-stand test in patients with multiple sclerosis.

DETAILED DESCRIPTION:
The population of the research will be participants with multiple sclerosis. The 30-second sit-to-stand test will be performed in the participant's home environment. . Patients will be instructed to cross their arms over their chest and complete as many standing cycles as possible in 30 seconds, standing until fully upright and then sitting until the hips touch the chair without the assistance of the hands. Inter-rater reliability will be assessed by two different raters in the same video interview. In contrast, intra-rater reliability will be evaluated by analyzing the number of repetitions recorded by the same rater in two different video interviews conducted 24-28 hours apart.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with MS according to the McDonald criteria by a neurologist
* having and being able to use a device with Internet access (e.g. smartphone, computer or tablet)
* having EDSS between 1.5 and 6.5,
* being between the ages of 18-65.

Exclusion Criteria:

* Patients who have had a recurrence of the disease in the last 30 days,
* have an additional health problem (orthopedic, neurological, internal or cardiorespiratory) that prevents standing/walking,
* do not agree to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: multiple sclerosis patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-03-11 (Estimated); Primary Completion 2024-06-24 (Estimated); Study Completion 2024-06-29 (Estimated)

PRIMARY OUTCOMES:
30 second sit and stand test | 24-48 hours
  The 30-second sit-to-stand test is a test used to evaluate lower extremity muscle strength, balance and walking functions.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu talu, Study Director — Inonu University

IPD SHARING:
Plan to Share IPD: Yes
Study data can be shared with other researchers if desired
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the study was published
Access Criteria: If requested from the authors, it can be shared with researchers at the authors' discretion.